CLINICAL TRIAL: NCT03499249
Title: A Phase 2 Trial of N-Acetylcysteine in Biliary Atresia After Kasai Portoenterostomy
Brief Title: N-Acetylcysteine in Biliary Atresia After Kasai Portoenterostomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sanjiv Harpavat, Assistant Professor, Department of Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-40962; 135796 (Other: FDA IND Identifier)
Record Dates: First submitted 2018-04-04; First posted 2018-04-17 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; N-Acetylcysteine; Glutathione; Kasai portoenterostomy; Bile flow; Serum bile acids; Serum bilirubin
MeSH Terms: conditions — Biliary Atresia | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This is a Phase 2 clinical trial using the two-stage "minimax" design described by Simon (Simon, 1989). As a Phase 2 trial, the trial's objective is to determine whether NAC has sufficient biological activity as adjunctive therapy for BA to warrant further study. By choosing the two-stage "minimax" design, we gain two advantages: (i) early termination if the drug is not efficacious, and (ii) using historical controls and therefore an overall smaller sample size to test the hypothesis, i.e., no randomization or control arm. This study design only identifies large effects (response >20%). For BA this is appropriate, because the field is in need of a robust therapy that can substantially limit liver damage and delay/prevent need for liver transplantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N-Acetylcysteine Treatment (Experimental): Will receive continuous intravenous NAC therapy (6.25 mg/kg/hour of 10 mg/ml solution, or 0.625 ml/kg/hour, to give 150 mg/kg/day), starting within 24 hours of completion of KP and lasting for a total of 7 days
  Interventions: Drug: N-Acetyl cysteine

INTERVENTIONS:
Drug: N-Acetyl cysteine — Intravenous NAC therapy (6.25 mg/kg/hour of 10 mg/ml solution, or 0.625 ml/kg/hour, to give 150 mg/kg/day), starting within 24 hours of completion of KP and lasting for a total of 7 days

SUMMARY:
Biliary atresia (BA) is a devastating liver disease of infancy, characterized by bile duct obstruction leading to liver fibrosis, cirrhosis, and eventual need for transplantation in most cases. BA is treated with Kasai portoenterostomy (KP). KPs can achieve bile drainage and improve outcomes. However, even with standard evidence of "good bile flow," bile flow rarely normalizes completely and liver disease continues to progress.

In this study, the investigators test whether intravenous N-acetylcysteine (NAC) can improve bile flow after KP. The rationale is that NAC leads to synthesis of glutathione, which is a powerful stimulator of bile flow. The primary objective is to determine whether NAC normalizes total serum bile acid (TSBA) concentrations within 24 weeks of KP. Achieving normal TSBAs is uncommon with current standard-of-care, and is predicted to be associated with better long-term outcomes. The secondary objectives are to describe how other parameters commonly followed in BA change with NAC therapy, as well as report adverse events occurring with therapy and in the first two years of life. This study follows the "minimax" Phase 2 clinical trial design.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a disease characterized by fibro-obliteration of extrahepatic bile ducts leading to impaired bile flow (Sokol et al., 2007). BA is treated with the Kasai portoenterostomy (KP), an operation which connects the liver directly to the intestine in attempt to relieve bile back-up and promote bile flow. KPs have variable success. KPs occasionally normalize bile flow and stop disease progression (Jimenez-Rivera et al., 2013). More commonly, however, bile flow never completely normalizes after KP. This can be detected by elevated total bilirubin (TB) or conjugated bilirubin (Bc) serum concentrations, or, when TB and Bc are normal, elevated total serum bile acids (TSBA) concentrations (Bezerra et al., 2014; Shneider et al., 2015; Venkat et al., 2014). Impaired flow leads to fibrosis, cirrhosis, and eventual need for liver transplantation. Given these uneven results, therapies are urgently needed to enhance the KP's success.

The investigators hypothesize that N-acetylcysteine (NAC) will improve outcomes after KP, because NAC is a precursor for the powerful choleretic molecule glutathione (Ballatori and Truong, 1989, 1992, Ballatori et al., 1986, 1989). The hypothesis assumes that better bile flow will lead to better outcomes. This is supported by previous reports demonstrating that good bile flow correlates with slower disease progression in BA. For example, a recent study showed infants with good bile flow after KP were significantly less likely to develop failure-to-thrive, ascites, hypoalbuminemia, or coagulopathy in the first two years of life (Shneider et al., 2015). Furthermore, these infants had significantly higher transplant-free survival in the same time period. In this study, TB <2.0 mg/dL within three months of KP was used as the marker for good bile flow.

NAC has a number of properties that make it an especially attractive potential therapeutic agent. First, glutathione creates an osmotic gradient in the bile duct lumen which drives one-third of total bile flow in humans (the other drivers are bile acids and secretin/bicarbonate) (Ballatori and Truong, 1989, 1992, Ballatori et al., 1986, 1989). Second, NAC is a Food and Drug Administration-approved therapy for another serious liver condition in neonates and children (acetaminophen overdose). It has also been used for other liver and non-liver indications in neonates, with few reported adverse events (Ahola et al., 2003; Flynn et al., 2003; Jenkins et al., 2016; Kortsalioudaki et al., 2008; Mager et al., 2008; Soghier and Brion, 2006; Squires et al., 2013; Wiest et al., 2014). Third, glutathione is an anti-oxidant, which could scavenge the free radicals contributing to cirrhosis. Preclinical studies are also promising, with glutathione's strong choleretic properties best established in rat flow studies and NAC's hepatoprotective effects documented in rescuing different mouse models of cholestasis (Ballatori et al., 1986; Galicia-Moreno et al., 2009, 2012; Tahan et al., 2007).

To test the hypotheses, the investigators will administer intravenous NAC continuously for seven days and determine the number of subjects with normal TSBAs (0-10 umol/L) within 24 weeks of KP. In addition, markers of BA progression, such as abnormal laboratory results, failure-to-thrive, and occurrence of complications related to chronic liver disease, will be described over the first two years of life. Finally, all adverse events occurring during NAC infusion and in the 21 days after its completion will be recorded. The study employs the two-stage "minimax" Phase 2 clinical trial design, a design commonly used in oncological trials to determine whether a particularly therapy has sufficient activity to warrant a larger Phase 3 trial (Simon, 1989). The two-stage "minimax" design offers two distinct advantages compared to other designs: (i) early termination if the drug is not efficacious; and (ii) small sample sizes, because historical controls rather than a separate control arm are used.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than or equal to 90 days at time of KP (standard age range in which KPs are performed)
2. BA diagnosis made by intraoperative cholangiography and KP performed at Texas Children's Hospital, Texas Medical Center Campus
3. Legal guardian(s) sign consent after understanding risks and investigational nature of study

Exclusion Criteria:

1. Decompensated liver disease (INR >1.3) despite parenteral Vitamin K administration)
2. KP not performed for any reason (i.e., normal intraoperative cholangiography, or liver found to be too diseased intraoperatively to proceed with KP)
3. Active respiratory infection
4. Renal impairment, as defined by having an eGFR < 60 mL/min/1.73m2 or creatinine clearance < 60 mL/min (https://www.niddk.nih.gov/health-information/communication-programs/nkdep/laboratory-evaluation/glomerular-filtration-rate-calculators/children-conventional-units)
5. Presence of severe concurrent illnesses, such as pulmonary (i.e., bronchopulmonary dysplasia), neurological, cardiovascular, metabolic, endocrine, and renal disorders, which may be congenital or acquired, that would interfere with the conduct and results of the study

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Harpavat, MD. PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital and Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahola T, Lapatto R, Raivio KO, Selander B, Stigson L, Jonsson B, Jonsbo F, Esberg G, Stovring S, Kjartansson S, Stiris T, Lossius K, Virkola K, Fellman V. N-acetylcysteine does not prevent bronchopulmonary dysplasia in immature infants: a randomized controlled trial. J Pediatr. 2003 Dec;143(6):713-9. doi: 10.1067/S0022-3476(03)00419-0. PMID 14657813
- [Background] Ballatori N, Truong AT. Relation between biliary glutathione excretion and bile acid-independent bile flow. Am J Physiol. 1989 Jan;256(1 Pt 1):G22-30. doi: 10.1152/ajpgi.1989.256.1.G22. PMID 2912148
- [Background] Ballatori N, Truong AT. Glutathione as a primary osmotic driving force in hepatic bile formation. Am J Physiol. 1992 Nov;263(5 Pt 1):G617-24. doi: 10.1152/ajpgi.1992.263.5.G617. PMID 1443136
- [Background] Ballatori N, Jacob R, Boyer JL. Intrabiliary glutathione hydrolysis. A source of glutamate in bile. J Biol Chem. 1986 Jun 15;261(17):7860-5. PMID 2872220
- [Background] Ballatori N, Truong AT, Ma AK, Boyer JL. Determinants of glutathione efflux and biliary GSH/GSSG ratio in perfused rat liver. Am J Physiol. 1989 Mar;256(3 Pt 1):G482-90. doi: 10.1152/ajpgi.1989.256.3.G482. PMID 2564253
- [Background] Bezerra JA, Spino C, Magee JC, Shneider BL, Rosenthal P, Wang KS, Erlichman J, Haber B, Hertel PM, Karpen SJ, Kerkar N, Loomes KM, Molleston JP, Murray KF, Romero R, Schwarz KB, Shepherd R, Suchy FJ, Turmelle YP, Whitington PF, Moore J, Sherker AH, Robuck PR, Sokol RJ; Childhood Liver Disease Research and Education Network (ChiLDREN). Use of corticosteroids after hepatoportoenterostomy for bile drainage in infants with biliary atresia: the START randomized clinical trial. JAMA. 2014 May 7;311(17):1750-9. doi: 10.1001/jama.2014.2623. PMID 24794368
- [Background] Flynn DM, Mohan N, McKiernan P, Beath S, Buckels J, Mayer D, Kelly DA. Progress in treatment and outcome for children with neonatal haemochromatosis. Arch Dis Child Fetal Neonatal Ed. 2003 Mar;88(2):F124-7. doi: 10.1136/fn.88.2.f124. PMID 12598501
- [Background] Galicia-Moreno M, Rodriguez-Rivera A, Reyes-Gordillo K, Segovia J, Shibayama M, Tsutsumi V, Vergara P, Moreno MG, Muriel P. N-acetylcysteine prevents carbon tetrachloride-induced liver cirrhosis: role of liver transforming growth factor-beta and oxidative stress. Eur J Gastroenterol Hepatol. 2009 Aug;21(8):908-14. doi: 10.1097/MEG.0b013e32831f1f3a. PMID 19398917
- [Background] Galicia-Moreno M, Favari L, Muriel P. Antifibrotic and antioxidant effects of N-acetylcysteine in an experimental cholestatic model. Eur J Gastroenterol Hepatol. 2012 Feb;24(2):179-85. doi: 10.1097/MEG.0b013e32834f3123. PMID 22241216
- [Background] Jenkins DD, Wiest DB, Mulvihill DM, Hlavacek AM, Majstoravich SJ, Brown TR, Taylor JJ, Buckley JR, Turner RP, Rollins LG, Bentzley JP, Hope KE, Barbour AB, Lowe DW, Martin RH, Chang EY. Fetal and Neonatal Effects of N-Acetylcysteine When Used for Neuroprotection in Maternal Chorioamnionitis. J Pediatr. 2016 Jan;168:67-76.e6. doi: 10.1016/j.jpeds.2015.09.076. Epub 2015 Nov 3. PMID 26545726
- [Background] Jimenez-Rivera C, Jolin-Dahel KS, Fortinsky KJ, Gozdyra P, Benchimol EI. International incidence and outcomes of biliary atresia. J Pediatr Gastroenterol Nutr. 2013 Apr;56(4):344-54. doi: 10.1097/MPG.0b013e318282a913. PMID 23263590
- [Background] Kortsalioudaki C, Taylor RM, Cheeseman P, Bansal S, Mieli-Vergani G, Dhawan A. Safety and efficacy of N-acetylcysteine in children with non-acetaminophen-induced acute liver failure. Liver Transpl. 2008 Jan;14(1):25-30. doi: 10.1002/lt.21246. PMID 18161828
- [Background] Lynch RM, Robertson R. Anaphylactoid reactions to intravenous N-acetylcysteine: a prospective case controlled study. Accid Emerg Nurs. 2004 Jan;12(1):10-5. doi: 10.1016/j.aaen.2003.07.001. PMID 14700565
- [Background] Mager DR, Marcon M, Wales P, Pencharz PB. Use of N-acetyl cysteine for the treatment of parenteral nutrition-induced liver disease in children receiving home parenteral nutrition. J Pediatr Gastroenterol Nutr. 2008 Feb;46(2):220-3. doi: 10.1097/MPG.0b013e3180653ce6. No abstract available. PMID 18223385
- [Background] Shneider BL, Magee JC, Karpen SJ, Rand EB, Narkewicz MR, Bass LM, Schwarz K, Whitington PF, Bezerra JA, Kerkar N, Haber B, Rosenthal P, Turmelle YP, Molleston JP, Murray KF, Ng VL, Wang KS, Romero R, Squires RH, Arnon R, Sherker AH, Moore J, Ye W, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Total Serum Bilirubin within 3 Months of Hepatoportoenterostomy Predicts Short-Term Outcomes in Biliary Atresia. J Pediatr. 2016 Mar;170:211-7.e1-2. doi: 10.1016/j.jpeds.2015.11.058. Epub 2015 Dec 24. PMID 26725209
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Soghier LM, Brion LP. Cysteine, cystine or N-acetylcysteine supplementation in parenterally fed neonates. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD004869. doi: 10.1002/14651858.CD004869.pub2. PMID 17054219
- [Background] Sokol RJ, Shepherd RW, Superina R, Bezerra JA, Robuck P, Hoofnagle JH. Screening and outcomes in biliary atresia: summary of a National Institutes of Health workshop. Hepatology. 2007 Aug;46(2):566-81. doi: 10.1002/hep.21790. PMID 17661405
- [Background] Squires RH, Dhawan A, Alonso E, Narkewicz MR, Shneider BL, Rodriguez-Baez N, Olio DD, Karpen S, Bucuvalas J, Lobritto S, Rand E, Rosenthal P, Horslen S, Ng V, Subbarao G, Kerkar N, Rudnick D, Lopez MJ, Schwarz K, Romero R, Elisofon S, Doo E, Robuck PR, Lawlor S, Belle SH; Pediatric Acute Liver Failure Study Group. Intravenous N-acetylcysteine in pediatric patients with nonacetaminophen acute liver failure: a placebo-controlled clinical trial. Hepatology. 2013 Apr;57(4):1542-9. doi: 10.1002/hep.26001. Epub 2013 Feb 4. PMID 22886633
- [Background] Tahan G, Tarcin O, Tahan V, Eren F, Gedik N, Sahan E, Biberoglu N, Guzel S, Bozbas A, Tozun N, Yucel O. The effects of N-acetylcysteine on bile duct ligation-induced liver fibrosis in rats. Dig Dis Sci. 2007 Dec;52(12):3348-54. doi: 10.1007/s10620-006-9717-9. Epub 2007 Apr 12. PMID 17436097
- [Background] Venkat VL, Shneider BL, Magee JC, Turmelle Y, Arnon R, Bezerra JA, Hertel PM, Karpen SJ, Kerkar N, Loomes KM, Molleston J, Murray KF, Ng VL, Raghunathan T, Rosenthal P, Schwartz K, Sherker AH, Sokol RJ, Teckman J, Wang K, Whitington PF, Heubi JE; Childhood Liver Disease Research and Education Network. Total serum bilirubin predicts fat-soluble vitamin deficiency better than serum bile acids in infants with biliary atresia. J Pediatr Gastroenterol Nutr. 2014 Dec;59(6):702-7. doi: 10.1097/MPG.0000000000000547. PMID 25419594
- [Background] Wiest DB, Chang E, Fanning D, Garner S, Cox T, Jenkins DD. Antenatal pharmacokinetics and placental transfer of N-acetylcysteine in chorioamnionitis for fetal neuroprotection. J Pediatr. 2014 Oct;165(4):672-7.e2. doi: 10.1016/j.jpeds.2014.06.044. Epub 2014 Jul 23. PMID 25064164
- [Derived] Harpavat S, Borovsky KA, Scheurer ME, Cavallo L, Erhiawarie FE, Vasudevan S, Vogel AM, Cerminara D, Tessier EM, Patel KR, Devaraj S, Shneider BL. A phase 2 trial of short-term intravenous N-acetylcysteine in biliary atresia after Kasai portoenterostomy. Hepatol Commun. 2025 Jun 9;9(7):e0729. doi: 10.1097/HC9.0000000000000729. eCollection 2025 Jul 1. PMID 40489761

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-Acetylcysteine Treatment
Started | 13
Completed | 12
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | N-Acetylcysteine Treatment
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 36 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic, all races | 7
  Non-Hispanic Asian | 1
  Non-Hispanic Black | 3
  non-Hispanic White | 2
Region of Enrollment [Number; unit: participants]
  United States | 13
Aspartate aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-glutamyltransferase (GGT) [Mean (Standard Deviation); unit: IU/L]
  AST | 123 (83)
  ALT | 80 (56)
  GGT | 360 (322)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Biliary Atresia (BA) Achieving Total Serum Bile Acids Less Than or Equal to 10 *U*Mol/L Within 24 Weeks of Kasai Portoenterostomy (KP)
Description: Expected is ~5% of participants based on historical controls (see protocol for summary of historical controls); a higher number is a better outcome
Time Frame: Within 24 weeks after KP
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetylcysteine Treatment
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-glutamyltransferase (GGT) Fold, and Conjugated Bilirubin (Bc) Change Above Baseline at 3 Days and 7 Days After KP (During Treatment)
Description: fold-change from baseline (ratio); a fold-change <1 is a better outcome.
Time Frame: 3 days after KP compared to baseline (before KP); 7 days after KP compared to baseline (before KP)
Measure: Mean (Standard Deviation); unit: fold change over baseline
Arm/Group | N-Acetylcysteine Treatment
Number analyzed (Participants) | 12
fold change over baseline
  AST 3 days after KP | 1.5 (0.5)
  AST 7 days after KP | 1.4 (0.4)
  ALT 3 days after KP | 3.3 (2.3)
  ALT 7 days after KP | 2.1 (0.5)
  GGT 3 days after KP | 0.9 (0.3)
  GGT 7 days after KP | 1.7 (0.9)
  Bc 3 days after KP | 1.3 (0.4)
  Bc 7 days after KP | 1.3 (0.4)

3. Secondary Outcome: Number of Patients Experiencing Sentinel Events in the First 2 Years of Life
Description: Events include Nasogastric (NG) feeds or Total Parental Nutrition (TPN) initiation, Splenomegaly (based on ultrasound findings), Thrombocytopenia (platelets <150,000/mm3), Ascites (recorded when diuretics were needed for fluid accumulation), GI bleed (varices documented by endoscopy), Portal hypertension (one of the following: ascites, or combination of splenomegaly and thrombocytopenia), and Liver transplant or death; units are number of patients, higher numbers are worse outcomes.
Time Frame: First two years of life
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetylcysteine Treatment
Number analyzed (Participants) | 12
Participants
  NG feeds or TPN initiation | 4
  Splenomegaly | 7
  Thrombocytopenia | 5
  Ascites | 4
  GI bleed | 0
  Portal hypertension | 5
  Liver transplant or death | 4

4. Secondary Outcome: Number of Patients With Adverse Events Possibly Related to NAC, Including Rash, Urticaria, Pruritus, Tachycardia, Hypotension, Vomiting, Edema, Anaphylaxis, and Intravenous Line Issues
Description: Units are number of patients, higher number is worse outcome
Time Frame: Within four weeks after KP
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetylcysteine Treatment
Number analyzed (Participants) | 13
Participants
  Tachycardia | 1
  Other | 0

ADVERSE EVENTS:
Time Frame: Within 28 days of KP (7 days of treatment and 21 days afterwards) for Serious adverse events, and Non-serious adverse events. Outcome measure. In first 2 years of life for All-Cause Mortality (this was also outcome measure #3).
Description: Non-serious: Emesis with feeds, Loss of an intravenous (IV) line, Febrile illness, AST 400 IU/L >pre-KP value, GGT 400 IU/L >pre-KP value, Conjugated bilirubin 3 mg/dL >pre-KP value, Total bilirubin 5 mg/dL >pre-KP value Serious: Febrile illness, ALT 700 IU/L >pre-KP value, INR >2.0, Tachycardia
Arm/Group | N-Acetylcysteine Treatment
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine Treatment (N=13)
Febrile illness (Infections and infestations) | 2 (2)
ALT 700 IU/L >pre-KP value (Hepatobiliary disorders) | 1 (1)
INR >2.0 (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine Treatment (N=13)
Emesis with feeds (Gastrointestinal disorders) | 3 (3)
Loss of an IV (Investigations) | 4 (4)
Febrile illness (Infections and infestations) | 1 (1)
AST 400 IU/L >pre-KP value (Hepatobiliary disorders) | 6 (6)
GGT 400 IU/L >pre-KP value (Hepatobiliary disorders) | 8 (8)
Conjugated bilirubin 3 mg/dL >pre-KP value (Hepatobiliary disorders) | 2 (2)
Total bilirubin 5 mg/dL >pre-KP value (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT03499249/Prot_SAP_000.pdf